CLINICAL TRIAL: NCT04412759
Title: PORCINE XENOGRAFT OR MICROBIAL CELLULOSE IN THE TREATMENT OF PARTIAL THICKNESS BURNS - A RANDOMISED CLINICAL TRIAL
Brief Title: PORCINE XENOGRAFT OR MICROBIAL CELLULOSE IN THE TREATMENT OF PARTIAL THICKNESS BURNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Folke Sjoberg, Professor in burn care, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC-2015
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Burns; Burn Scar; Burn Second Degree
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Porcine xenograft (No Intervention): porcine xenograft derived from dermal porcine skin. Standard of care treatement for partila thickness burn at the specfic centre
- Microbial cellulose (Experimental): Novel dressing consisting of a biopolymer spun by the bacteria Acetobacter xylinum (later removed).
  Interventions: Other: microbial cellulose

INTERVENTIONS:
Other: microbial cellulose — polymer dressing synthesized in abundance with Acetobacter Xylinum
  Arms: Microbial cellulose

SUMMARY:
The purpose of this study was to compare two wound dressing products for partial thickness burns in adults.

DETAILED DESCRIPTION:
After being informed about the study, all patients that had given written informed consent underwent screening. If eligible study participants were randomized to be treated wih either the standard dressing of care; pigskin or a microbial cellulose. Dressing were applied within 72 hours after burn injury. Evaluation was done in an open manner due to the specific characteristics of the dressings. Study particpants were followed weekly until complete wound closure and after that evaluated at 6 and 12 months after injruy for burn scar outcome.

ELIGIBILITY:
Inclusion Criteria:

* Study participants admitted within 72 hours of injury
* partial-thickness burns requiring a temporary skin cover
* written informed consent

Exclusion Criteria:

* severe coexisting cutaneous trauma
* chronic or current skin disease,
* severe cognitive dysfunction or psychiatric disorder
* pregnant or breast feeding women were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Time to complete healing of the burn | Evaluated at each visit (1-3 times per week) from admission until complete healing, up to 6 months
  Healing time was calculated from the date of injury to the date when the wound bed was assessed as completely (100 %) re-epithelialized, with no need for further dressing changes other than protection against shearing according to the treating physician.

SECONDARY OUTCOMES:
Burn wound infection | Evaluated at each visit (1-3 times per week) from admission until complete healing, up to 6 months
  Wound infections were diagnosed (by the burn surgeon) if they fulfilled at least two of the following criteria:
  (based on the American Burn Association definition of burn wound infection)
  * Clinical signs such as localised pain and swelling, spreading erythema, and heat at the affected site.
  * Positive bacterial culture growth of the surface wound swab.
  * Signs of systemic infection indicated by a rise in CRP concentration (reference range < 10 mg/L for capillary sampling) together with increased body temperature where other sources of infection have been excluded.
Burn wound pain | Evaluated at each visit (1-3 times per week) from admission until complete healing, up to 6 months
  The patients were asked to estimate the burn wound pain at rest, during activity, and during dressing changes using a numerical rating scale (NRS) where 0 indicated no pain and 10 the worst pain ever imaginable.
Duration of hospital stay (LOS) | From admission until discharge, up to 6 months
  All patients hospitalized for their burns were monitored by the study nurse and the day of discharge was noted in the CRF. Any readmission after initial discharge was also noted and included in the total length of stay.
Burn scar outcome | Evaluated at six and 12 months after injury
  Burn scar outcome was evaluated using the Patient Observer Scar Assessment Scale (POSAS). The scale includes two separate subscales, The Observer Sscale, used by an experienced burn occupational therapist and the Patient Sscale, used by the study participants.

CONTACTS AND LOCATIONS:
Locations (1):
- The Burn Centre at Linköping University Hospital,, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No